CLINICAL TRIAL: NCT05610293
Title: Tumor Free Survival in T1 Squamous Cell Carcinomas of the Lip Treated With 5mm or 10mm Surgical Margins.
Brief Title: T1 Squamous Cell Carcinomas of the Lip
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-2224-A-2
Record Dates: First submitted 2022-11-02; First posted 2022-11-09 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Lip; Lip Cancer; Lip SCC; Squamous Cell Carcinoma; Squamous Cell Carcinoma of the Lip; Surgery; Surgical Margin; Recurrence; Metastasis; Tumor Free Margins
Keywords: Disease free survival; Multicenter; Histological margin
MeSH Terms: conditions — Lymphoid Interstitial Pneumonia; Lip Neoplasms; Carcinoma, Squamous Cell; Margins of Excision; Recurrence; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 5mm surgical margin: Patients treated with a 5mm surgical margin for a T1 SCC of the lip.
- 10mm surgical margin: Patients treated with a 10mm surgical margin for a T1 SCC of the lip.

SUMMARY:
The purpose of this study is to investigate the risk of recurrence and metastasis in patients treated with different surgical margins (5mm vs 10mm) for a T1 squamous cell carcinoma of the lip.

DETAILED DESCRIPTION:
The incidence of head and neck tumors, including lip carcinomas, in increasing. Exact incidences are lacking because in the Dutch National Cancer Registry (NCR) lip carcinomas are registered both as oral cavity carcinomas and skin carcinomas. In 2021, 136 patients with lip cancer were registered in the Netherlands. 90% of patients with lip cancer have localized disease (stage 1) with a 5-year survival rate of more than 90%.

Lip carcinomas usually involve squamous cell carcinomas (SCC). In most cases, the SCC is located on the sun-exposed lower lip. In approximately 90% of lower lip SCCs, the tumor is smaller than 2cm in diameter. According to the current eight edition of the Tumor Node Metastasis (TNM) classification of the American Joint Committee on Cancer (AJCC) and the ninth edition of the Union for Internation Cancer Control (UICC), it is classified as tumor stage I.

Surgery is the conventional treatment for a T1 SCC of the lip, where tumor margins can be verified via histologic examination. A histologic margin of less than 2mm is associated with an increased risk of local recurrence and metastasis.

In the Netherlands, surgical treatment of lip carcinomas is performed by dermatologists, plastic and reconstruction surgeons, oral and maxillofacial surgeons (OMFS), and otorhinolaryngologists (ENT). There is currently no international consensus regarding the appropriate surgical margins for excision of a T1 SCC on the lip. According to the AJCC, a surgical margin of 5mm is appropriate, while according to the UICC, a surgical margin of 10mm is appropriate. Scientific evidence is limited regarding differences in tumor clearance and the risk of recurrence or metastasis after excision of T1 SCCs with a surgical margin of 5mm versus 10mm.

We aimed to investigate whether there is a significant difference in tumor-free survival in patients with surgically treated T1 lip SCC with a surgical margin of 5mm versus 10mm.

A retrospective descriptive multicenter data study will be conducted with four different centers in the Netherlands (Maastricht University Medical Center+), Radboud University Medical Center (RadboudUMC) Nijmegen, Catharina Hospital Eindhoven (CZE), and Zuyderland Medical Center Heerlen/Sittard. Data will be obtained from the Dutch Cancer Registry (NKR) and the Dutch Pathological Anatomical National Automated Archive (PALGA).

The primary outcome is the difference in tumor-free survival in patients treated with surgical margins of 5mm and 10mm. The secondary outcome is the difference in tumor-free survival in patients with different histologic free margins. To evaluate the risk of surgical and histologic margins on the risk of local recurrence and metastasis, a Kaplan-Meier analysis, log-rank test and cox-proportional hazard models will be used.

ELIGIBILITY:
Inclusion Criteria:

* patients of 18 years and older
* with a T1 cutaneous squamous cell carcinoma of the lip (including the cutaneous lip, vermillion border, vermillion and mucosal involvement).
* who received surgical treatment
* treated at one of the following centers: Maastricht University Medical Center+ (MUMC+), Radboud University Medical Center (Radboudumc), Zuyderland Medical Center (Zuyderland MC), Catharina Hospital Eindhoven (CZE).

Exclusion Criteria:

* malignancies other than cutaneous squamous cell carcinoma
* Oropharyngeal cancer
* patients with stage T2-T4 cutaneous squamous cell caricnomas of the lip

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data from patients are collected retrospectively using data from the Pathological Anatomical National Automated Archive (PALGA). These are data from patients treated at one of the following four centers in the Netherlands: MUMC+, Radboudumc, Zuyderland MC, CZE.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Tumor-free survival surgical margins | 5 years after surgical treatment
  Difference in tumor-free survival of patients treated with a 5mm surgical margin versus 10mm surgical margin for a T1 SCC on the lip. An event was refered to as the occurrence of recurrence or metastasis.

SECONDARY OUTCOMES:
Tumor-free survival histologic margins | 5 years after surgical treatment
  Difference in tumor-free survival of patients with a histologic margin of <2mm versus patients with a histologic margin of 2mm or more of their T1 SCC on the lip.

CONTACTS AND LOCATIONS:
Overall Officials: K Mosterd, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (3):
- Netherlands (3):
  - Radboud UMC, Nijmegen, Gelderland
  - Catharina Hospital, Eindhoven
  - Zuyderland Medical Center, Heerlen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kerawala C, Roques T, Jeannon JP, Bisase B. Oral cavity and lip cancer: United Kingdom National Multidisciplinary Guidelines. J Laryngol Otol. 2016 May;130(S2):S83-S89. doi: 10.1017/S0022215116000499. PMID 27841120
- [Background] de Visscher JG, Grond AJ, Botke G, van der Waal I. Results of radiotherapy for squamous cell carcinoma of the vermilion border of the lower lip. A retrospective analysis of 108 patients. Radiother Oncol. 1996 Apr;39(1):9-14. doi: 10.1016/0167-8140(96)01716-1. PMID 8735488
- [Background] Kelleners-Smeets NW, Bekkenk MW, de Haas ER. [Skin cancer: from smearing to cutting]. Ned Tijdschr Geneeskd. 2013;157(12):A5602. Dutch. PMID 23515035
- [Background] Biasoli ER, Valente VB, Mantovan B, Collado FU, Neto SC, Sundefeld ML, Miyahara GI, Bernabe DG. Lip Cancer: A Clinicopathological Study and Treatment Outcomes in a 25-Year Experience. J Oral Maxillofac Surg. 2016 Jul;74(7):1360-7. doi: 10.1016/j.joms.2016.01.041. Epub 2016 Jan 30. PMID 26917204
- [Background] de Visscher JG, Gooris PJ, Vermey A, Roodenburg JL. Surgical margins for resection of squamous cell carcinoma of the lower lip. Int J Oral Maxillofac Surg. 2002 Apr;31(2):154-7. doi: 10.1054/ijom.2002.0232. PMID 12102412
- [Background] Joo YH, Cho JK, Koo BS, Kwon M, Kwon SK, Kwon SY, Kim MS, Kim JK, Kim H, Nam I, Roh JL, Park YM, Park IS, Park JJ, Shin SC, Ahn SH, Won S, Ryu CH, Yoon TM, Lee G, Lee DY, Lee MC, Lee JK, Lee JC, Lim JY, Chang JW, Jang JY, Chung MK, Jung YS, Cho JG, Choi YS, Choi JS, Lee GH, Chung PS. Guidelines for the Surgical Management of Oral Cancer: Korean Society of Thyroid-Head and Neck Surgery. Clin Exp Otorhinolaryngol. 2019 May;12(2):107-144. doi: 10.21053/ceo.2018.01816. Epub 2019 Feb 2. PMID 30703871
- [Background] O'Sullivan B. UICC manual of clinical oncology: John Wiley & Sons; 2015.
- See also: Integral cancer center Netherlands; incidence rates on lip tumors — https://iknl.nl/nkr-cijfers